CLINICAL TRIAL: NCT06302673
Title: The Role Of Laserpuncture For Prevention Of Nausea And Vomiting Post Strabismus Surgery With General Anesthesia In Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yossie Faudina Putri, doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23081229
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial (RCT)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laserpuncture (Experimental): Laserpuncture : using RJ Laser with Nogier B wave setting, frequency 584 Hz, power 50 mW, wavelength 785 nm, and energy of 2 Joules at each acupuncture point ( PC6 Neiguan and CV12 Zhongwan)
  Interventions: Device: Laserpuncture
- Sham-Laserpuncture (Sham Comparator): Sham Laserpuncture: The laser is turned on but not activated at each acupuncture point ( PC6 Neiguan and CV12 Zhongwan)
  Interventions: Device: Sham Laserpuncture

INTERVENTIONS:
Device: Laserpuncture — Laserpuncture : using RJ Laser with Nogier B wave setting, frequency 584 Hz, power 50 mW, wavelength 785 nm, and energy of 2 Joules at each acupuncture point ( PC6 Neiguan and CV12 Zhongwan)
  Arms: Laserpuncture
Device: Sham Laserpuncture — Sham Laserpuncture: The laser is turned on but not activated at each acupuncture point ( PC6 Neiguan and CV12 Zhongwan).
  Arms: Sham-Laserpuncture

SUMMARY:
This study to determine the effectiveness of a combination of pre-surgical laserpuncture with standard anti-emetic therapy for PONV symptoms in adult patients after strabismus surgery under general anesthesia compared to a combination of pre-surgical placebo laserpuncture with standard anti-emetic therapy. Research design using a double blinded randomized controlled trial (RCT) where research subjects and data takers who will be disguised. The research will be carried out in the Operation and Inpatient Room, Kirana Building, RSUPN Dr. Cipto Mangunkusumo (RSCM) with research subjects as adult patients undergoing strabismus surgery under general anesthesia. Assessment of nausea and vomiting using AVS ( Analog Visual Scale) consists of scoring using a score from 1-5 which indicates the severity of nausea and vomiting.

DETAILED DESCRIPTION:
This clinical trial is to evaluate the role of laserpuncture as a prevention of nausea and vomiting in adult patients after strabismus surgery under general anesthesia. Participants are 32 males/females aged 18-59 years. They will be divided into 2 groups: (1) Group laserpuncture and (2) Sham laserpuncture. The study intervention was performed 30 minutes before surgery. The primary outcome in this study was the incidence of postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18-59 years.
2. Patients undergoing simple strabismus surgery involving no more than two muscles without transposition under general anesthesia.
3. Meets the ASA (American Society of Anesthesiologists) score of 1-2.
4. Complete the surgical preparations according to the presedation sheet.
5. Sign the informed consent sheet.
6. Patients who can communicate with the research team.
7. Patients undergoing surgery <3 hours.

Exclusion Criteria:

1. The patient is pregnant.
2. Patients who have a history of drug or drug abuse.
3. Patients with hypersensitivity to laser light.
4. There are wounds or skin disorders at the radiation site (skin TB, SLE(Systemic Lupus Erythematosus) skin
5. Patients who have gastrointestinal diseases (intestinal obstruction, peristaltic disorders gastrointestinal tract, gastroenteritis, irritable bowel syndrome, dyspepsia,gastroesophageal reflux disease/GERD, appendicitis, hepatitis, cholecystitis, inflammatory bowel synchrome, pancreatitis, peptic ulcer, peritonitis, food poisoning).
6. Patients with metabolic diseases (acid-base imbalance, metabolic diseases calcium, glucose metabolism disease, hyperlactemia, mitochondrial disease, phenylketonuria)
7. Patients with conditions of high intracranial pressure, head trauma, migraines, disease with symptoms of seizures, vestibular diseases, malignancies, mental and psychogenic diseases, diseases arising from consumption of drugs, nephrolithiasis, other kidney diseases, myocardial infarction, as well as the occurrence of nausea and vomiting before surgery.
8. Infection accompanied by high fever (temperature >38°C)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Analog Visual Scale for nausea vomitting | 30 minutes after surgery, 2 hours after surgery, 6 hours after surgery, and 12 hours after surgery.
  PONV (post operative nausea vomiting) assessment based on the onset of nausea
  * vomit that has value 1-5. 1 = No nausea and vomiting. 2 = Nausea and possible vomiting tolerated, with the nausea episode can't remember by the patient or intensity nausea low with one vomiting episodes (not needed antiemetic additional inside both events). Ordinal 57 3 = Nausea and vomiting, with episodes that don't can be remembered and need antiemetic. 4 = Nausea and possible vomiting remembered clearly and need antiemetic for control symptom. 5=Nausea and persistent vomiting, with nothing symptom improvement even if given antiemetic.

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia - Cipto Mangunkusumo Hospital
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No